CLINICAL TRIAL: NCT01338064
Title: Oxidative Stress Biomarkers to Monitor and Early Detect Health Impairment in Workers Exposed to Silica (Caesar Stone)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Elizabeth Fairman, Tel Aviv medical center
Other Study IDs: TASMC-11-YS-619-CTIL
Record Dates: First submitted 2011-02-06; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Silicosis
Keywords: Silicosis
MeSH Terms: conditions — Silicosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Induced sputum (IS)
  2. Exhaled Breath Condensate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- exposed workers: At least six months of occupational exposure to Caesar stone

SUMMARY:
Silicosis is well-known occupational disease caused by free crystalline silica (silicon dioxide) and is marked by inflammation and pulmonary fibrosis. There are cumulative evidences that exposure to Caesar stone (quartz surface products that manufactured from up to 93% quartz, polymer resins and pigments) is particularly dangerous to exposed workers.

Goals: To examine marble workers exposed to Caesar Stone in order to propose a working plan of surveillance and prevention by biological monitoring.

DETAILED DESCRIPTION:
Study participants would be recruited during two years of the study. They will be asked to come to a single visit at Pulmonary Laboratory of Tel Aviv Medical Center. During the meeting, participants will be given a precise explanation about the tests they will perform and after signing the informed consent will perform following tests:

1. Induced sputum (IS) - will be done after pretreatment with short acting beta-2 agonist and 3% saline will be administrated by an ultrasonic nebulizer for up to 20 min. Differential cell count, particle size distribution test of the particulate matter (with a Eyetech Analyzer (Ankersmid, Yokneam, Israel)will be done from IS samples and evaluation the activity of Heme oxygenase 1 (HO-1) protein from IS supernatants.
2. EBC-Exhaled Breath Condensate-will be done by condensation expiratory air and particulate matter and markers of oxidation will be measured.
3. Participants will be asked to complete occupational questionnaire.
4. Pulmonary function tests (PFTs): The measurement will be performed using standard protocols according to American Thoracic Society/European Respiratory Society (ATS/ERS) guidelines. Including Lung diffusion testing.

Laboratory tests of induced sputum and EBC will be done within a week of a participant visit. Analysis of data will be done after the completion of data collection and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. male
2. 18-70 years old
3. At least six months of professional exposure to Caesar stone

Exclusion Criteria:

1. Other occupational exposure (welding of any kind)
2. Chronic Obstructive Pulmonary Disease (COPD), tuberculosis, asthma, autoimmune disease in healthy exposed workers
3. Interstitial lung disease in exposed workers with clinically approved silicosis

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least six months of occupational exposure to Caesar stone
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite silicosis according to ATS/ERS guidelines | one day
  1. Occupational physician examination
  2. Pulmonary function tests (PFTs): The measurement will be performed using standard protocols according to ARS/ERS guidelines. Including Lung diffusion testing
  3. Computed Tomography (CT) test if need

SECONDARY OUTCOMES:
Particle size distribution of the particulate matter | one day
  Particle size distribution test of the particulate matter (with a Eyetech Analyzer (Ankersmid, Yokneam, Israel) will be done from Induced sputum (IS) samples and EBC-Exhaled Breath Condensate.
The activity of Heme oxygenase 1 (HO-1) protein | one day
  Evaluation the activity of Heme oxygenase 1 (HO-1) protein will be done from Induced sputum (IS) supernatants.
Differential cell count | one day
  Differential cell count will be done from Induced sputum (IS) samples.
Markers of oxidation | one day
  Markers of oxidation will be measured will be measured in EBC-Exhaled Breath Condensate.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Shwartz, MD, Principal Investigator — Tel Aviv medical center. Pulmonary and Allergy department
Locations (1):
- Pulmonary Laboratory of Tel Aviv Sourasky Medical Center, Tel Aviv, Israel